CLINICAL TRIAL: NCT01485003
Title: A Multicenter, Observational, Open-Label, Single-Arm Study of Tysabri in Early Relapsing-Remitting Multiple Sclerosis in Anti-JCV Antibody Negative Patients
Brief Title: Observational Study of Tysabri in Early Relapsing-Remitting Multiple Sclerosis in Anti-JC Virus Antibody Negative Participants
Acronym: STRIVE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 101MS407
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Biological: natalizumab — Natalizumab will not be provided as a part of this study. Participants will receive natalizumab as prescribed by their treating physician.
  Other Names: BG00002; Tysabri

SUMMARY:
The primary objective of the study is to determine which baseline and yearly response factors (clinical and para clinical) predict overall disease-free status at Month 12 and Month 24, and clinical disease-free status in subsequent Months 36 and 48. The secondary objectives are: To identify prognostic factors at Baseline that predict overall disease-free status at Month 12, and to assess if yearly overall disease-free response factors predict overall disease-free status at Month 24; To evaluate clinical disease-free status (relapse, Expanded Disability Status Scale [EDSS]) at each analysis time point of Months 12, 24, 36, and 48; To identify prognostic factors at Baseline that predict clinical disease-free status at Month 12, and to assess yearly clinical disease-free response factors that predict clinical disease-free status (relapse, EDSS) in subsequent years at Months 24, 36, and 48; To evaluate the impact of Tysabri at each analysis time point of Months 12, 24, 36, and 48 on the following: annualized relapse rate (ARR), sustained EDSS progression and improvement (24-week sustained); To evaluate the impact of Tysabri at each analysis time point of Months 12, 24, 36, and 48 on the following: magnetic resonance image (MRI) measures: T2, T1, T1 with Gadolinium (Gd), brain atrophy; To evaluate the impact of Tysabri at Month 24 and Month 48 on the following: optical coherence tomography (OCT), Low and High Contrast Visual Acuity Assessment; To evaluate the impact of Tysabri at each analysis time point of Months 12, 24, 36, and 48 on the following: cognitive impairment (Symbol Digit Modalities Test [SDMT]), capacity for work (Work Productivity and Activity Impairment Questionnaire [WPAI]), quality of life (QoL) (Multiple Sclerosis Impact Scale [MSIS-29])

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of Relapsing Multiple Sclerosis (McDonald 2010 Criteria ).
* <3 year disease duration.
* Must have an Expanded Disability Status Scale (EDSS) score from 0 to 4.0, inclusive.
* Anti-JCV antibody negative test within 6 months of Screening Visit.
* Must satisfy the approved therapeutic indications for Tysabri.
* Must be treatment-naïve to disease-modifying therapy (DMT) or have been treated with DMT (including but not limited to Avonex, Betaseron, Rebif, Copaxone, Extavia, or Gilenya) for ≤36 months total prior to date of informed consent.
* Decision to treat with Tysabri must precede enrollment.

Key Exclusion Criteria:

* Any prior treatment with Tysabri.
* Anti-JCV antibody positive at any timepoint prior to the Screening Visit.
* Contraindications to treatment with Tysabri as described in the US Prescribing Information.
* History of progressive multifocal leukoencephalopathy (PML) or other opportunistic infections, or an increased risk for such infections.
* History of diagnosis of Primary Progressive Multiple Sclerosis (PPM) and/or Secondary Progressive Multiple Sclerosis (SPMS).
* Receiving immunomodulatory or immunosuppressive therapy.
* Prior history of immunosuppressive use (mitoxantrone, azathioprine, methotrexate, cyclophosphamide, mycophenolate, cladribine, rituximab).
* Immunocompromised at the time of enrollment.
* Known active malignancies (subjects with cutaneous basal cell carcinoma that has been completely excised prior to study entry remain eligible).
* Women breastfeeding, pregnant, or planning to become pregnant; women who are not post-menopausal or surgically sterile who are unwilling to practice contraception.
* Inability to comply with study requirements.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited by participating neurologists from among their MS patients who opt to begin treatment with Tysabri.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants who are overall disease activity-free at Months 12 and 24 | Baseline and Months 12 and 24
  Overall disease activity-free is defined as no relapses, no disability progression (RRMS), and absence of MRI disease activity (no gadolinium [gd])+ lesions, no new or enlarging T2-hyperintense lesions). A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. Sustained disability progression defined by at least a 1.0-point increase on the EDSS from a Baseline EDSS ≥1.0 that is sustained for 12 or 24 weeks, or at least a 1.5-point increase on the EDSS from a Baseline EDSS <1.0 that is sustained for 12 or 24 weeks. The EDSS measures the disability status of people with multiple sclerosis on a scale that ranges from 0 to 10, with higher scores indicating more disability.
Proportion of participants who are clinical disease activity-free at Months 36 and 48 | Baseline and Months 36 and 48
  Clinical disease activity-free is defined as no sustained EDSS progression and no relapses at Month 36 and 48.

SECONDARY OUTCOMES:
Identification of baseline prognostic factors that predict overall disease-free status | Baseline and Month 12
Identification of yearly overall disease-free response factors that predict overall disease-free status | Month 12 and Month 24
Number of Participants with Clinical Disease-Free Status Measured by Relapses | Months 12, 24, 36, and 48
  A clinical relapse is a new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement.
Identification of baseline prognostic factors that predict clinical disease-free status | Month 12
Identification of yearly clinical disease-free response factors that predict clinical disease-free status | Months 24, 36 and 48
Annualized Relapse Rate | Months 12, 24, 36, and 48
  A clinical relapse is defined as new or recurrent neurological symptoms, not associated with fever, lasting for at least 24 hours, and followed by a period of 30 days of stability or improvement. The ARR will be calculated by tabulating the total number of relapses experienced in the group divided by the number of days up to the end of study, and the ratio then multiplied by 365.
Percentage of participants with Sustained EDSS progression | Baseline and Months 12, 24, 36, and 48
Sustained EDSS improvement | Baseline and Months 12, 24, 36, and 48
  Sustained improvement in disability is defined as participants with Baseline EDSS of at least 2.0 who experience a ≥1.0 decrease in EDSS that is sustained for 24 weeks.
Change form baseline in number of new or newly enlarging T2 hyperintense lesions as assessed by MRI | Baseline and Months 12, 24, 36, and 48
Change from baseline in number of new T1 hypointense lesions as assessed by MRI | Baseline and Months 12, 24, 36, and 48
Change form baseline in number of T1 lesions with Gd-enhancing lesions as assessed by MRI | Baseline and Months 12, 24, 36, and 48
MRI brain atrophy as assessed by MRI | Baseline and Months 12, 24, 36, and 48
Change from baseline in retinal nerve fiber layer (RNFL) thickness as assessed by OCT | Baseline and Month 24 and Month 48
Change from baseline in low contrast visual acuity | Baseline and Month 24 and Month 48
  Low-contrast visual acuity testing captures the minimum size at which individuals can perceive letters of a particular contrast level (shade of gray on white background). Using the low-contrast Sloan letter charts at 2.5% and 1.25% low contrast levels, participants will be asked to read each of the 2 charts at a 2-meter distance using a standardized testing protocol.
Change from baseline in high contrast visual acuity | Baseline and Month 24 and Month 48
  High contrast acuity testing is important to help determine the smallest letters a person can read on a standardized visual acuity chart or on a card held 14 - 20 feet away. A visual acuity test is a routine part of an eye examination.
Cognitive impairment as assessed by change from baseline in SDMT | Baseline and Months 12, 24, 36 and 48
  SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best).
Capacity for work as assessed by change from baseline in WPAI questionnaire | Baseline and Months 12, 24, 36 and 48
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteeism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Quality of Life as measured by MSIS-29 | Baseline and Months 12, 24, 36 and 48
  The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a participant-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a participant's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health.
Number of Participants with Clinical Disease-Free Status Measured by EDSS | Months 12, 24, 36 and 48
  Expanded Disability Status Scale (EDSS) is a method of quantifying disability in 8 Functional Systems (FS) and allows neurologists to assign a Functional System Score (FSS) in each of these. The FSS include pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral (or mental), and other. Each of the FSS is an ordinal clinical rating scale ranging from 0 to 5 or 6, with higher scores indicating more disability. These ratings are then used in conjunction with observations and information concerning gait and use of assistive devices to rate the EDSS. The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments. Each of the FSS and the EDSS are single-item scales and there is no composite or summed score.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (42):
- United States (42):
  - Research Site, Homewood, Alabama
  - Research Site, Sun City, Arizona
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Fort Collins, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Wellesley Hills, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, East Lansing, Michigan
  - Research Site, Lincoln, Nebraska
  - Research Site, Freehold, New Jersey
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Plainview, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Gahanna, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington

REFERENCES:
- [Derived] Perumal J, Balabanov R, Balcer L, Galetta S, Sun Z, Li H, Rutledge D, Avila RL, Fox RJ. Long-Term Effectiveness and Safety of Natalizumab in African American and Hispanic/Latino Patients with Early Relapsing-Remitting Multiple Sclerosis: STRIVE Data Analysis. Neurol Ther. 2023 Jun;12(3):833-848. doi: 10.1007/s40120-023-00461-0. Epub 2023 Mar 26. PMID 36966440
- [Derived] Perumal J, Balabanov R, Su R, Chang R, Balcer LJ, Galetta SL, Avila RL, Rutledge D, Fox RJ. Correction to: Improvements in Cognitive Processing Speed, Disability, and Patient-Reported Outcomes in Patients with Early Relapsing-Remitting Multiple Sclerosis Treated with Natalizumab: Results of a 4-year, Real-World, Open-Label Study. CNS Drugs. 2023 Mar;37(3):275-289. doi: 10.1007/s40263-022-00982-6. PMID 36780107
- [Derived] Perumal J, Balabanov R, Su R, Chang R, Balcer LJ, Galetta SL, Avila RL, Rutledge D, Fox RJ. Improvements in Cognitive Processing Speed, Disability, and Patient-Reported Outcomes in Patients with Early Relapsing-Remitting Multiple Sclerosis Treated with Natalizumab: Results of a 4-year, Real-World, Open-Label Study. CNS Drugs. 2022 Sep;36(9):977-993. doi: 10.1007/s40263-022-00950-0. Epub 2022 Sep 5. PMID 36064841
- [Derived] Perumal J, Balabanov R, Su R, Chang R, Balcer L, Galetta S, Campagnolo DI, Avila R, Lee L, Rutledge D, Fox RJ. Natalizumab in Early Relapsing-Remitting Multiple Sclerosis: A 4-Year, Open-Label Study. Adv Ther. 2021 Jul;38(7):3724-3742. doi: 10.1007/s12325-021-01722-w. Epub 2021 May 20. PMID 34014549
- [Derived] Perumal J, Fox RJ, Balabanov R, Balcer LJ, Galetta S, Makh S, Santra S, Hotermans C, Lee L. Outcomes of natalizumab treatment within 3 years of relapsing-remitting multiple sclerosis diagnosis: a prespecified 2-year interim analysis of STRIVE. BMC Neurol. 2019 Jun 8;19(1):116. doi: 10.1186/s12883-019-1337-z. PMID 31176355